CLINICAL TRIAL: NCT06114186
Title: FAM (Follower, Action Plan, and Remote Monitoring) Intervention to Reduce Severe Hyperglycemia in Adults With Type 1 Diabetes Mellitus at Risk for Diabetic Ketoacidosis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MED-2023-32321
Record Dates: First submitted 2023-10-16; First posted 2023-11-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: randomized 1:1 to the intervention or control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- control group (Active Comparator): anticipate 8 CGM and 2 non-CGM user dyads in the control group
  Interventions: Device: FAM intervention consisting of a Follower of glucose data, Action Plan, and Remote Monitoring of glucose data
- intervention group (Experimental): anticipate 8 CGM and 2 non-CGM user dyads in the intervention group
  Interventions: Other: standard of care

INTERVENTIONS:
Device: FAM intervention consisting of a Follower of glucose data, Action Plan, and Remote Monitoring of glucose data — using remote monitoring and real-time glucose data sharing with a Follower.
  Arms: control group
Other: standard of care — self reported HbA1C or GMI
  Arms: intervention group

SUMMARY:
Diabetic ketoacidosis (DKA) results in significant morbidity and healthcare utilization and is the main contributor to loss of life expectancy in people with diabetes mellitus type 1 (T1DM) <50 years old. This suggests the need to develop interventions to reduce DKA events. Innovative features of newer continuous glucose monitoring devices offer opportunities for novel strategies to reduce DKA. Designating a family member, friend, or caregiver as a Follower was associated with reduction in HbA1C, increased time in range, and improvement in quality of life metrics in people with T1DM. However, the previously published studies are limited as they were either retrospective, survey-based, or do not overlap with our proposed cohort involving adults ages 18-65 with T1DM (prior prospective studies involved either pregnant women with T1DM or adults ≥60 years of age with T1DM). This study is a randomized controlled trial pilot study to evaluate an intervention (FAM) using a Follower, Action Plan, and Remote Monitoring of glucose data to reduce severe hyperglycemia, a modifiable risk factor for DKA, in adults with T1DM at high risk for DKA. The intervention uses real-time glucose data sharing with a Follower (family member, friend, or caregiver) and personalized diabetes education provided to the dyad (person with T1DM and their chosen Follower). The overall hypothesis is that the FAM intervention will improve glycemia with the primary outcome studied in this preliminary pilot study being percentage of time spent with glucose ≥250 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* People with T1DM for ≥1 year ages 18 - 65
* HbA1C ≥7.5.0% - 14.0%
* If the person with T1DM uses a CGM, the CGM must have the capability of real-time data sharing including glycemic alerts with a Follower (including but not limited to Dexcom G6 or G7 or FreeStyle Libre 2 or 3, or Medtronic Guardian Sensor 3)
* Follower (family member or friend ages 18 years and older) willing to participate in the study and "follow" glucose data and who was no self-reported cognitive impairment
* Ability of the dyad (participant and Follower) to communicate and provide consent in English
* CGM users: ≥50% personal CGM use and ≥50% Dexcom G6 Pro CGM use during the pre-intervention period (days -14 to -1)
* Non CGM users: ≥50% Dexcom G6 Pro CGM use and average ≥2 BGM readings/day during the pre-intervention period (days -14 to -1)

Exclusion Criteria:

* Prisoner
* Active treatment with a sodium-glucose cotransporter-2 inhibitor or planning to start a sodium-glucose cotransporter-2 inhibitor in the next 6 months
* Active malignancy with the exception of non-melanoma skin cancer
* Hospice
* Skin conditions that inhibit wearing a CGM sensor and known severe allergy to adhesives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
percentage of time with severe hyperglycemia | 90 days
  number of continuous glucose monitoring or blood glucose monitoring readings with glucose ≥250 mg/dL divided by the total number of readings

SECONDARY OUTCOMES:
Hyperglycemia - Continuous Glucose Monitor glucose monitor (CGM) metrics | 90 days
  -Percentage of time glucose >180 mg/dL
Severe hyperglycemia >400 mg/dL - Continuous Glucose Monitor glucose monitor (CGM) metrics | 90 days
  -Percentage of time glucose >400 mg/dL
Hypoglycemia - continuous glucose monitor | 90 days
  -Percentage of time glucose< 70 mg/dL
Hemoglobin A1c | days 0 and 90
  -HbA1c
Level 2 Hypoglycemia - Continuous Glucose Monitor | 90 days
  -Percentage of time glucose < 54 mg/dL
Time in Range - Continuous Glucose Monitor | 90 days
  -Percentage of time glucose is 70 - 180 mg/dL
Glycemic variability - Continuous Glucose Monitor | 90 days
  -Glycemic variability
Glucose Management Indicator - Continuous Glucose Monitor | 90 days
  -Glucose Management Indicator
Number of glucose reading/day - Blood Glucose Monitor | 90 days
  -Number of glucose readings/day
Hyperglycemia - Blood Glucose Monitor | 90 days
  -Percentage of time glucose <180 mg/dL
Severe Hyperglycemia > 400 mg/dL - Blood Glucose Monitor | 90 days
  -Percentage of time glucose >400 mg/dL
Hypoglycemia - Blood Glucose Monitor | 90 days
  -Percentage of time glucose< 70 mg/dL
Level 2 Hypoglycemia -Blood Glucose Monitor | 90 days
  -Percentage of time glucose < 54 mg/dL
Time in Range - Blood Glucose Monitor | 90 days
  -Percentage of time glucose is 70 - 180 mg/dL
Ketone assessment | 90 days
  -Frequency and severity of ketonuria assessed using urine ketone test strips
Assessment of the intervention's efficacy and its burden on participants | 90 days
  -Questionnaire
Hypoglycemic Confidence Scale | 90 days
  * Likert Scale
  * Minimum value: Not Confident At All
  * Maximum value: Very Confident
Diabetes Distress Scale for Adults with T1DM | 90 days
  * Likert Scale
  * Minimum value: A Very Serious Problem
  * Maximum value: Not a Problem
Diabetes Empowerment Scale | 90 days
  * Likert Scale
  * Minimum value: Strongly Disagree
  * Maximum value: Strongly Agree
36-Item Short-Form Health Survey | 90 days
  -Questionnaire
Hypoglycemic Confidence Scale for Partners of Adults with T1DM | 90 days
  * Likert Scale
  * Minimum value: Not Confident At All
  * Maximum value: Very Confident
Diabetes Distress Scale for Partners of Adults with T1DM | 90 days
  * Likert Scale
  * Minimum value: A great deal
  * Maximum value: Not at all

OTHER OUTCOMES:
Hospitalization for DKA | 90 days
  -The number of DKA-related hospitalizations for each participant will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kohlenberg, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States